CLINICAL TRIAL: NCT01008384
Title: The Effect of Vitamin D Repletion on Small LDL Particle Number in Subjects at Elevated Cardiovascular Risk
Brief Title: The Effect of Vitamin D Repletion on Small Low Density Lipoprotein (LDL) Particle Number in Subjects at Elevated Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: MAP-0683
Record Dates: First submitted 2009-10-22; First posted 2009-11-05 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (No Intervention)
- Vitamin D3 (Experimental): Vitamin D3 given for 8 weeks
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 50,000 units taken orally once a week for 8 weeks
  Arms: Vitamin D3

SUMMARY:
Vitamin D is a fat-soluble vitamin that is naturally present in very few foods, added to others, and available as a dietary supplement. It is also produced in the body when ultraviolet rays from sunlight strike the skin and trigger vitamin D synthesis. Vitamin D is essential for promoting calcium absorption and maintaining adequate serum calcium and phosphate concentrations to enable normal mineralization of bone and bone growth. Without sufficient vitamin D, bones can become thin, brittle, or misshapen. Vitamin D sufficiency prevents rickets in children and osteomalacia in adults. Together with calcium, vitamin D also helps protect older adults from osteoporosis. Many people have low levels of Vitamin D. Replacing Vitamin D is thought to help lower the risk of heart disease. Vitamin D may be helpful, but it could also be harmful. The investigators are studying the effect of Vitamin D on the level of a harmful kind of cholesterol. Participants will have their cholesterol levels measured and then receive either Vitamin D or a placebo. After 2 months of treatment, the investigators will measure their cholesterol levels again.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years and < 85 years
2. Vitamin D 25-OH level <20 ng/ml
3. One of the following risk factors:

   * Known coronary artery disease (CAD) or a CAD equivalent (e.g. diabetes, chronic kidney disease, etc)
   * BMI > 30 kg/m2
   * Random Glucose Level > 200mg/dl
   * Increased Waist Circumference (male: > 40in; Females: > 35in.)
   * Decreased HDL (Male: < 40mg/dl; Female: < 50mf/dl)
   * Framingham Risk Score > 10%
   * hsCRP > 2 mg/L

Exclusion Criteria:

1. Serum phosphorus level > 5.5 mg/dl
2. Estimated GFR <30 ml/min/1.73m2
3. Use of Vitamin D >400 IU/day within 1 month of most recent Vitamin D 25-OH determination
4. Use of calcitriol or other "activated" vitamin D
5. Change in statin, ezetimibe, niacin, fibrate dose within 1 month
6. Concurrent participation in an investigational drug study
7. Have any other condition, which in the opinion of the investigator, should prohibit the participation in the study
8. Serum calcium level >10.5 mg/dl
9. anti-epileptic medication
10. triglycerides > 400 mg/dL
11. BMI > 40 kg/m2
12. Evidence of cirrhosis as evidenced by AST > 3 x upper limit, ALT > 3 x upper limit, bilirubin > 1.5 mg/dL , albumin < 3.0 g/dL, PT > 14.5 sec
13. Pregnant or Lactating Females

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Small LDL particle concentration | Visit 5

CONTACTS AND LOCATIONS:
Overall Officials: Manish Ponda, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

REFERENCES:
- [Derived] Ponda MP, Dowd K, Finkielstein D, Holt PR, Breslow JL. The short-term effects of vitamin D repletion on cholesterol: a randomized, placebo-controlled trial. Arterioscler Thromb Vasc Biol. 2012 Oct;32(10):2510-5. doi: 10.1161/ATVBAHA.112.254110. Epub 2012 Sep 4. PMID 22947589